CLINICAL TRIAL: NCT04633668
Title: Pilot RCT of the Impact of Cognitive Behavioral Therapy on Parasomnias
Brief Title: Impact of Cognitive Behavioral Therapy on Parasomnias
Acronym: parasomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Nora Vincent, Psychologist/Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Umanitoba1
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Parasomnia
MeSH Terms: conditions — Parasomnias | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: 2 (group) X 3 (time)
Who Masked: Participant
Masking Description: Self-Monitoring of sleep
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-p (Experimental): cognitive behavioral therapy, Monitoring of sleep through sleep diaries, nightmare experiences, and actigraphy
  Interventions: Behavioral: CBT for parasomnias (CBT-p)
- Self-monitoring (Active Comparator): Monitoring of sleep through sleep diaries, nightmare experiences, and actigraphy
  Interventions: Behavioral: Self-Monitoring

INTERVENTIONS:
Behavioral: CBT for parasomnias (CBT-p) — Psychoeducation, sleep hygiene, imagery re-scripting, scheduled awakenings, safety planning, cognitive therapy, and stress management for 6 weeks
  Arms: CBT-p
Behavioral: Self-Monitoring — Monitoring of sleep quality through sleep diary, actigraphy, nightmare experiences for 6 weeks
  Arms: Self-monitoring

SUMMARY:
This research aims to determine whether cognitive behavioral therapy can effectively reduce parasomnias in a sample of 20 adult outpatients with Non-REM and REM parasomnias. A secondary objective is to assess whether treatment produces improvements in daytime energy, mood, and anxiety symptoms, as well as functional impairment (work/leisure activities).

DETAILED DESCRIPTION:
Sleep wake disorders are prevalent and impactful conditions often poorly assessed and sub-optimally treated in the clinical setting. Undiagnosed sleep disorders can masquerade as mental health conditions and worsen the outcomes associated with these conditions. Further, sleep disorders can develop from mental health conditions and the reverse is also true (particularly for mood disorders). Successful treatment of sleep disorders requires a targeted approach.

Parasomnias are unwanted physical or mental events that occur during sleep or during arousal from sleep. The states of wakefulness, NREM, and REM are normally distinct and occur in an organized and predictable pattern over the 24-hour period. However, in parasomnias, aspects of more than one state co-occur and intermix. There are four types of parasomnias identified by the Diagnostic and Statistical Manual of Mental Disorders ( DSM 5). These include two NREM parasomnias: sleepwalking and sleep terrors, and two REM parasomnias: nightmare disorder and REM sleep behaviour disorder (RSBD). Lifetime prevalence of these conditions ranges from 6.9% (sleepwalking) to 67% (nightmare disorder).

In general, NREM parasomnia events are primed by conditions that increase sleep pressure and triggered by sleep-disrupting factors. They are more likely to occur following sleep restriction or deprivation, when SWS rebounds. Immediate triggers of sleepwalking in adults are sleep disruptions associated with sleep-disordered breathing, periodic limb movements, noises and touch. Pilon et al. induced episodes in adult sleepwalkers, but not in non-sleepwalkers, with specific auditory stimuli and this effect was accentuated under conditions of prior sleep deprivation.

Currently accepted interventions for parasomnias include pharmacological and psychological treatments. Pharmacological interventions involve the use of sedating medications (benzodiazepines, tricyclic antidepressants) or alpha-1 blocker (Prazosin).

Cognitive Behavioral Therapy. Psychological treatments primarily rely on cognitive behavioral therapy to achieve better sleep hygiene, reduced hyperarousal, and to teach the ability to practice with reducing cognitive arousal during the sleep period through planned rehearsal and scheduled awakenings. There are no well elaborated and systematic treatment packages for Non-REM parasomnias and so this protocol will represent an innovation in this area. Therefore, the purpose of the study is to develop and test such a package.

Self-Monitoring of Sleep. Self-monitoring of disturbed sleep has been shown to produce small but significant positive impacts on some aspects of sleep (e.g., insomnia). As there is no widely accepted placebo for parasomnia treatment, this is viewed as an adequate control condition.

Objectives This research aims to determine whether cognitive behavioral therapy can effectively reduce parasomnias in a sample of 20 adult outpatients with Non-REM and REM parasomnias. A secondary objective is to assess whether treatment produces improvements in daytime energy, mood, and anxiety symptoms, as well as functional impairment (work/leisure activities). The hypotheses of the study are that participants who receive a 6-week program CBT-p therapy will report fewer episodes of parasomnia than those who self-monitor their sleep for 6 weeks, and will have objectively better sleep as measured by the prodigy and actigraphy at one-week (T2) post treatment and at two months post treatment (T3).

METHODS Trial Design This will be a single-blind randomized controlled trial with two conditions.

ELIGIBILITY:
Inclusion Criteria:

* DSM 5 Parasomnia Disorder
* at least one parasomnia event per week
* daytime fatigue or sleepiness
* 6 months in duration

Exclusion Criteria:

* current use of agents known to triggers parasomnias such as Lithium carbonate, Thioridazine, Chlorpromazine, Perhphenazine, Methaqualone, or Amitriptyline,
* for participants taking benzodiazepines or Prazosin, a stable dose regime for the past 4 weeks,
* excessive alcohol consumption defined as the consumption of > 10 alcoholic beverages per week

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Parasomnia events | 6 weeks
  # of parasomnia events
Nocturnal Activity | 6 weeks
  activity level during sleep period
Nightmares | 6 weeks
  Nightmare Experiences Scale, 0-16, higher scores more problematic nightmares

SECONDARY OUTCOMES:
Fatigue | 6 weeks
  Multi-Dimensional Fatigue Inventory, 0-16, higher scores mean more fatigue
Sleepiness | 6 weeks
  Epworth Sleepiness Scale, 0-24, higher scores mean more sleepiness
Insomnia | 6 weeks
  Insomnia Severity Index, 0-28, with higher scores meaning more insomnia
Cognitive | 6 weeks
  PROMIS Applied Cognition Scale, 4-20, with higher scores meaning better cognition
Impairment | 6 weeks
  Work and Social Adjustment Scale, 0-40, higher scores mean more impairment
Depression, Anxiety, and Stress | 6 weeks
  Depression, Anxiety, and Stress Scale, o-63, with higher scores meaning more depression, anxiety, and stress

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Rempel-Rossum, Study Director — University of Manitoba
Locations (1):
- Psychealth Center, 771 Bannatyne Avenue, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vincent N, Dirkse D, Giannouli E, McQuarrie A. Transdiagnostic cognitive behavioral therapy for nightmares and parasomnias. J Clin Sleep Med. 2023 Mar 1;19(3):499-509. doi: 10.5664/jcsm.10374. PMID 36468650